CLINICAL TRIAL: NCT02687061
Title: Retrieval of Patients Chronically Infected With Hepatitis B or Hepatitis C in Northern Holland
Brief Title: Chronic Hepatitis B and C Recall Northern Holland
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Stichting MDL Holland-Noord (Other)
Collaborators: Gilead Sciences (Industry)
Responsible Party: Sponsor
Other Study IDs: NL-174-2008
Record Dates: First submitted 2016-02-08; First posted 2016-02-22 (Estimated); Last update posted 2016-02-22 (Estimated); Status verified 2016-02

CONDITIONS: Hepatitis B; Hepatitis C
Keywords: Recall study; Lost to follow-up
MeSH Terms: conditions — Hepatitis B; Hepatitis C

STUDY DESIGN:
Observational Model: Cohort
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Chronic hepatitis B: Patients diagnosed with chronic hepatitis B
- Chronic hepatitis C: Patients diagnosed with chronic hepatitis C

SUMMARY:
The project aims to retrieve patients diagnosed with chronic hepatitis B (cHB) and hepatitis C (cHC) who are lost to follow-up.Data files of the Public Health System and microbiology laboratories will be explored for registered cases of cHB and cHC. Subsequently the investigators will compare the registered cases with the list of known cHB and cHC patients in hospital care. Patients lost to follow up will be informed and approached via either the Public Health Service (PHS) or their primary care physician. Identified patients will be invited for re-evaluation at the regional hepatitis centre (The North Western Hospital, formerly Medical Centre Alkmaar) to assess the current status of their chronic disease. Evaluation will be performed in accordance with (inter-)national guidelines, no extra interventions will be performed.

After completion of re-evaluation, a final report will be made and send to both patient and primary care physician with recommendations for further follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of chronic hepatitis B (two positive HBsAg measurements with an interval of 6 months)
* Diagnosis of chronic hepatitis C (two positive anti-HCV with an interval of 6 months)

Exclusion Criteria:

* Already known in specialized care for chronic HBV or chronic HCV
* Cured from chronic HBV or chronic HCV

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The groups will be selected from registries of the Public Health Service (PHS) and medical microbiology laboratories. All positive anti-HCV and HBsAg will be checked and if patients with positive HBsAg or HCV are not known in specialised/hospital care, they will be included in our database.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2016-02; Primary Completion 2016-09 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Liver-related morbidity | Baseline
  At baseline, development of liver related morbidity due to chronic viral hepatitis will be assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Klemt-Kropp, MD, PhD, Principal Investigator — Stichting MDL Holland-Noord